CLINICAL TRIAL: NCT05076877
Title: A Phase 1, Open-label, Study in Healthy Participants to Evaluate the Effect of Steady State Concentrations of Lazertinib (JNJ-73841937) on the Single-dose Pharmacokinetics of Probe Substrates (Midazolam, Rosuvastatin, and Metformin)
Brief Title: A Study of Lazertinib (JNJ-73841937) in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR109080; 73841937NSC1008 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-09-17; First posted 2021-10-13 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Healthy
MeSH Terms: interventions — lazertinib; Midazolam; Rosuvastatin Calcium; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lazertinib + Probe Substrates of Midazolam, Rosuvastatin, and Metformin (Experimental): Participants will receive a single oral dose of probe substrates of midazolam, rosuvastatin, and metformin on Day 1 under fasted conditions followed by a single oral dose of lazertinib under fed conditions from Day 5 to Day 14 except Day 13 which is under fasted conditions and co-administered with probe substrates under fasted conditions on Day 13.
  Interventions: Drug: Lazertinib; Drug: Midazolam; Drug: Rosuvastatin; Drug: Metformin

INTERVENTIONS:
Drug: Lazertinib — Lazertinib tablets will be administered orally, alone or in combination with probe substrates.
  Other Names: JNJ-73841937; YH25448
Drug: Midazolam — Midazolam (cytochrome P450 3A4 [CYP3A4] substrate) will be administered orally as a syrup as a part of probe substrates.
Drug: Rosuvastatin — Rosuvastatin (breast cancer resistant protein [BCRP] substrate) tablet will be administered orally as a part of probe substrates.
Drug: Metformin — Metformin (organic cation transporter 1 [OCT1] substrate) will be administered orally as a syrup as a part of probe substrates.

SUMMARY:
The purpose of this study is to evaluate the effect of steady-state concentrations of lazertinib on the single-dose pharmacokinetics (PK) of probe substrates (midazolam, rosuvastatin, and metformin) in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of medical history at screening only, and physical examination, vital signs, and 12-lead electrocardiogram (ECG) performed at screening and at admission to the study center
* Healthy on the basis of clinical laboratory tests performed at screening and at admission to the study center.
* A woman who is considered surgically sterile but not postmenopausal, must have a negative highly sensitive serum (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test on Study Day 1. (exemptions: pregnancy test not required in female participants with prior hysterectomy or prior bilateral oophorectomy)
* Male participants must agree to use an adequate contraception method as deemed appropriate by the investigator
* Non-smoker or not using tobacco containing products for at least 6 months before first study drug administration and test negative for cotinine at screening and Study Day 1

Exclusion Criteria:

* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy, that in the opinion of the investigator, with written concurrence with the sponsor's medical monitor is considered cured with minimal risk of recurrence)
* History of suspected or confirmed coronavirus disease 2019 within 4 weeks before intake of study drug, or tests positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at admission to the study site
* Known allergies, hypersensitivity, or intolerance to lazertinib or its excipients or probe substrates
* Taken any disallowed therapies, concomitant therapy before the planned first dose of study drug
* Had major surgery, (example, requiring general anesthesia) within 8 weeks before screening, or will not have fully recovered from surgery, or has surgery planned during the time the participant is expected to participate in the study or within 4 weeks after the last dose of study drug administration

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Plasma Concentration of Probe Substrates (Midazolam, Rosuvastatin, and Metformin) Co-administered with Lazertinib (Day 13) as Test Versus Plasma Concentration of Probe Substrates Administered Alone (Day 1) as Reference | Predose up to 12 hours postdose (Days 1 and 13)
  Plasma samples will be analyzed to determine concentrations of midazolam and its metabolite 1-OH-midazolam, rosuvastatin, metformin, or lazertinib using a validated, specific, and sensitive method on Day 1 versus Day 13 as a part of drug-drug interaction (DDI) assessment.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 56 days
  AE is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with AEs by Severity | Up to 56 days
  Number of participants with AEs by severity will be reported. AE severity is a clinical determination of the intensity of an AE and is assessed by using the standard grades as follows: Grade 1= mild, Grade 2= moderate, Grade 3= severe, Grade 4= life-threatening and Grade 5= death related to AE.
Number of Participants with Clinically Significant Changes in Laboratory Test Results | Up to 28 days
  Number of participants with change in clinical laboratory test results (including hematology and serum chemistry) will be reported.
Number of Participants with Clinically Significant Abnormalities in 12-lead Electrocardiograms (ECGs) | Up to 28 days
  Number of participants with clinically significant abnormalities in ECGs will be reported.
Number of Participants with Clinically Significant Abnormalities in Vital Signs | Up to 28 days
  Number of participants with clinically significant abnormalities in vital signs (including temperature [oral], pulse rate, and blood pressure) will be reported.
Number of Participants with Clinically Significant Abnormalities in Physical Examination | Up to 28 days
  Number of participants with clinically significant abnormalities in physical examination (including height and body weight) will be reported.
Plasma Concentrations of Lazertinib at steady-state | Predose on Day 7, 9, 11, 13, and 14
  Plasma concentration of lazertinib at steady-state will be assessed.
Plasma Concentrations of Lazertinib Following Repeat Dosing for 10 Days | Day 14, 15, 16, 17, 21, and 28
  Plasma concentration of lazertinib following repeat dosing for 10 days will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency